CLINICAL TRIAL: NCT07032519
Title: Mindfulness Intervention for Fibromyalgia Delivered Through a Smartphone App
Acronym: Fibroapp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Asimina Lazaridou, PhD, Assistant Professor of Anesthesiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P001410
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
Keywords: Mindfulness; Pain; mHealth; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial utilizing a parallel assignment model. Participants are randomly assigned to either the intervention group, which receives a smartphone-based mindfulness video series and daily pain rating prompts, or a control group that receives daily pain tracking only. The intervention is self-guided and delivered remotely via a secure smartphone app. Outcomes are measured at baseline, post-intervention, and 3- and 6-month follow-ups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Intervention (MBI) (Experimental): Participants in this group will receive access to a smartphone app delivering an 8-week mindfulness-based intervention. The app includes weekly video modules (mindfulness practice and psychoeducation), daily pain tracking, and weekly assessments.
  Interventions: Behavioral: Mindfulness Intervention
- Control (No Intervention): Participants in this group will complete the same daily and weekly assessments via the smartphone app but will not have access to the mindfulness or psychoeducation content.

INTERVENTIONS:
Behavioral: Mindfulness Intervention — Participants will use the smartphone app daily for pain tracking and weekly to engage with mindfulness content and complete additional assessments.
  Arms: Mindfulness-Based Intervention (MBI)

SUMMARY:
The purpose of this pilot feasibility study is to evaluate the effects of a smartphone-based mindfulness intervention (MBI) on pain-related outcomes in individuals with fibromyalgia. This 8-week randomized controlled trial will compare an MBI app group to a control group who completes assessments only through the app.

The MBI intervention includes weekly video content focused on mindfulness practice and psychoeducation, combined with daily symptom tracking through the app. Participants in both groups will complete self-report measures at baseline, post-intervention, and follow-ups at 3 and 6 months.

The study will enroll up to 100 participants from Brigham and Women's Hospital and the greater Boston area. This pilot study is designed to assess feasibility and explore preliminary effects on outcomes such as pain interference, fibromyalgia symptoms, pain catastrophizing, sleep disturbance, emotional distress, mindfulness, and pain acceptance. Results will be used to inform the design of a future fully powered randomized trial.

DETAILED DESCRIPTION:
Mindfulness-based interventions have shown promise in improving symptoms of chronic pain, including fibromyalgia, through mechanisms such as increased pain acceptance, reduced catastrophizing, and enhanced emotional regulation. Delivering such interventions via smartphone application increases accessibility and scalability, particularly for individuals who face mobility or geographic barriers to in-person treatment.

This study uses a parallel-group randomized controlled design. Participants will be assigned to either the MBI intervention group or a control group. The intervention group will receive access to weekly mindfulness practice and psychoeducation videos through a smartphone app over the course of 8 weeks, in addition to daily symptom tracking and weekly assessments. The control group will use the same app to complete assessments only.

Primary outcomes include feasibility and clinical variables including pain interference, fibromyalgia symptoms, and pain catastrophizing. Secondary outcomes include sleep disturbance, anxiety, depression, pain acceptance, and mindfulness.

Assessments will be collected at baseline and after the 8-week intervention, with additional follow-ups at 3 and 6 months post-intervention to examine sustained effects. All study procedures, including informed consent, intervention delivery, and assessments, will occur remotely through the app or secure platforms.

The results of this study will offer insight into the acceptability, engagement, and preliminary efficacy of smartphone-based mindfulness interventions for fibromyalgia and guide development of a larger confirmatory trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65
* Diagnosis of fibromyalgia per Wolfe et al. (2011) criteria
* Stable medication regimen or medication-free
* Fluent in English
* Able to provide informed consent

Exclusion Criteria:

* Comorbid pain condition more severe than fibromyalgia
* Pregnancy or breastfeeding
* Current psychosis or history of severe psychiatric illness
* Active suicidal ideation
* Participation in another therapeutic trial
* Any condition that may interfere with study compliance as judged by the PI or study coordinator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Brief Pain Inventory | Daily for 8-weeks
  Assessed using the Brief Pain Inventory - Pain Interference Subscale

SECONDARY OUTCOMES:
Change in Fibromyalgia Symptoms (FIQR) | Weekly for 8-weeks
  Assessed using the Fibromyalgia Impact Questionnaire Revised
Change in Pain Catastrophizing (PCS) | Baseline and post (8 weeks)
  Assessed using the Fibromyalgia Impact Questionnaire Revised
Pain Acceptance (CPAQ-R) | Baseline and post (8 weeks)
  Assessed using the Chronic Pain Acceptance Questionnaire Revised
Mindfulness (MAAS) | Baseline and post (8 weeks)
  Assessed using the Mindful Attention Awareness Scale
Anxiety and Depression (PROMIS-A/D) | Baseline and post (8 weeks)
  Assessed using PROMIS Anxiety and Depression short forms
Qualitative Exit Interviews | Post (after 8-weeks)
  open-ended exit questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Asimina Lazaridou, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- The Brigham and Women's Hospital Department of Anesthesiology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No